CLINICAL TRIAL: NCT01723111
Title: A Prospective, Multicenter, Observational Study to Evaluate the Impact of Peritoneal Dialysis Compared With Hemodialysis on Iron Metabolism and Hepcidin
Brief Title: Impact of Dialysis Modality on Hepcidin and Iron Metabolism
Acronym: HERMES
Status: Completed | Type: Observational
Sponsor: Kyungpook National University Hospital (Other)
Collaborators: Roche Pharma AG (Industry); Fresenius Medical Care North America (Industry)
Responsible Party: Principal Investigator, Yong-Lim Kim, MD, PhD, Kyungpook National University Hospital
Other Study IDs: knuhhermes
Record Dates: First submitted 2012-11-02; First posted 2012-11-07 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: End-stage Renal Disease
Keywords: hepcidin; ESA; hemodialysis; peritoneal dialysis; iron metabolism; dialysis modality
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2 ml serum will be retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Peritoneal dialysis: start PD
- Hemodialysis: start HD

SUMMARY:
* Dialysis modality may influence the oxidative stress and proinflammatory cytokines in ESRD patients.
* Dialysis modality may affect hepcidin
* Dialysis modality may influence iron and ESA requirements.

DETAILED DESCRIPTION:
It has been considered that PD patients tended to be less anemic and require lower ESA dose than HD patients. In addition, it was also known that the level of oxidative stress and inflammatory cytokines tended to be lower in PD patients than HD patients. And hepcidin synthesis is markedly increased during inflammation. Altogether, Lower ESA requirement in PD patients may be associated with lower hepcidin level due to lower inflammatory state compared with HD patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18 years or older
* Dialysis treatment was expected over 3 months
* In HD patients, regular hemodialysis 4 h a session more than two times a week
* In PD patients, over 2 exchange with more than 1.5 L solution

Exclusion Criteria:

* Poorly controlled hypertension, i.e. sitting blood pressure exceeding 180/110 despite medication requiring hospitalization or interruption of ESA treatment
* Significant acute or chronic bleeding such as overt gastrointestinal bleeding within the previous 3 months
* Active malignant disease (except non-melanoma skin cancer and patients with malignant disease who have been disease-free for at least the 5 previous years are eligible)
* Acute infection
* Hemolysis
* Hemoglobinopathies (e.g. homozygous sickle-cell disease, thalassemia of all types)
* Megaloblastic anemia
* Platelet count >500 x 109/L or <100 x 109/L
* Pure red call aplasia
* Epileptic seizure during previous 3 months
* Women of childbearing potential without effective contraception
* Known hypersensitivity to recombinant human erythropoietin, polyethylene glycol
* Planned elective surgery during the study period except for cataract surgery or laser photocoagulation
* Life expectancy less than 12 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: New ESRD patients whose dialysis treatment is expected over 3 months
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-11; Primary Completion 2016-02 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
ESA (Erythrocyte stimulating agents) dose | six months
  We will compare ESA dose between PD patients and HD patients

SECONDARY OUTCOMES:
IV iron treatment (% of patients) | six months
  We will compare IV iron treatment (% of patients) between PD patients and HD patients
Hepcidin level | six months
  We will compare hepcidin level between PD patients and HD patients
hs-CRP | six months
  We will compare hs-CRP level between PD patients and HD patients
Myeloperoxidase | six months
  We will compare myeloperoxidase between PD patients and HD patients
Transfusion rate | six months
  We will compare transfusion rate ( % of patients) between PD patients and HD patients
TNF-a | six months
  We will compare TNF-a between PD patients and HD patients
IL-6 | six months
  We will compare IL-6 between PD patients and HD patients
Total antioxidant capacity | six months
  We will compare total antioxidant capacity between PD patients and HD patients

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Lim Kim, Principal Investigator — Division of Nephrology, Department of Internal Medicine, Kyungpook National University School of Medicine
Locations (4):
- South Korea (4):
  - Daegu Fatima Hospital, Daegu
  - Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University College of Medicine, Daegu

REFERENCES:
- [Background] Malyszko J, Malyszko JS, Kozminski P, Mysliwiec M. Type of renal replacement therapy and residual renal function may affect prohepcidin and hepcidin. Ren Fail. 2009;31(10):876-83. doi: 10.3109/08860220903216071. PMID 20030521